CLINICAL TRIAL: NCT03476096
Title: Sublingual Microcirculation Change in Pregnant Women With or Without High Risk Pregnancy Factors During Pregnancy and Postpartum Period
Brief Title: Sublingual Microcirculation Change During Pregnancy and Postpartum Period
Acronym: Cytocam-OBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201711067RINC
Record Dates: First submitted 2018-02-20; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-02

CONDITIONS: Microcirculation in Pregnancy
Keywords: pregnancy; microcirculation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control: healthy pregnant women
- Pre-eclampsia: high-risk pregnant women

SUMMARY:
Sublingual microcirculation change in pregnant women with or without high risk pregnancy factors during pregnancy and postpartum period.

DETAILED DESCRIPTION:
Microcirculation system is composed of a group of blood vessels less than 100 um in diameter composed of arterioles, capillaries, veins and other structures. The health of microcirculation system correlates well with the stability of systemic circulation. Perfusio of microcirculation is often affected by major diseases such as sepsis, shock and heart disease. Through various microcirculation monitoring instruments, the investigators can assess the disease severity and prognosis.

Physiological changes during pregnancy will increase the blood volume, stroke volume, and microcirculation. Preeclampsia refers to the development of hypertension (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg) after 20 weeks of gestation with proteinuria. Severe preeclampsia is associated with impaired endothelial cell circulation throughout the body, and reduced sublingual microcirculation perfusion.

Through the sublingual microcirculation monitor, studies have shown that pregnant women have more microcirculation perfusion than non-pregnant women, while women with severe preeclampsia and those with HELLP syndrome have impaired microcirculation.

This study aims to investigate whether there is any change in the sublingual microcirculation before and after labor in healthy pregnant women and high-risk pregnant women (such as epilepsy, gestational diabetes, etc.) through the third generation of microcirculation imaging microscope (cytocam).

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women older than 20 years old who will delivery baby in our hospital (both normal spontaneous delivery and cesarean section).
* Women over 20 years of age who will delivery baby in our hospital (both normal spontaneous delivery and cesarean section) and meet the definition of high-risk pregnancy such as gestational diabetes mellitus, placenta previa, placenta accreta, gestational hypertension, preeclampsia or severe preeclampsia.

Exclusion Criteria:

* Chronic hypertension or diabetes

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: healthy pregnant women and high-risk pregnant women (gestational diabetes mellitus, placenta previa, placenta accreta, gestational hypertension, preeclampsia or severe preeclampsia.)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes of perfused vessel density | From the day before delivery to three days after delivery
  Changes of perfused vessel density before and after delivery

SECONDARY OUTCOMES:
Changes of microvascular flow index | From the day before delivery to three days after delivery
  Changes of microvascular flow index before and after delivery
Changes of heterogeneity index before | From the day before delivery to three days after delivery
  Changes of heterogeneity index before and after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan